CLINICAL TRIAL: NCT05351905
Title: A Single-centre, Pilot, Randomized Controlled Trial of Oral Cannabinoids for Improving Pain Disability in Patients With Chronic Pain
Brief Title: Improving Pain Disability With the Use of Oral Cannabinoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Research Manager, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-5944
Record Dates: First submitted 2022-04-04; First posted 2022-04-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Opioid Use; Cannabis
MeSH Terms: conditions — Chronic Pain; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either a placebo, CBD oil (medical cannabis) or CBD+THC oil (medical cannabis) in a 1:1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, study staff, care providers, adjudicators, data analysts and investigators will be blinded to the active ingredient(s) in the study medication and group allocation. Blinding of all research team members who interact with the patient will avoid biases in communications with, or treatment of, participants based on group allocation. Blinding of research participants will avoid any bias in reporting (e.g., of pain ratings, side effects) and actions/behaviours during the study (e.g., opioid medication dose adjustments) based on group allocation and/or expectations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD oil (Experimental): Participants will receive CBD (cannabidiol) oil for a total duration of 12 weeks.
  Interventions: Drug: CBD oil ( MPL-001)
- CBD+THC oil (Experimental): Participants will receive CBD (cannabidiol) oil in combination with THC (delta-9-tetrahydrocannabinol) for a total duration of 12 weeks.
  Interventions: Drug: CDB+THC oil (MPL-005)
- Placebo oil (Placebo Comparator): Participants will receive matching placebo oil for a total duration of 12 weeks.
  Interventions: Drug: Placebo oil

INTERVENTIONS:
Drug: CBD oil ( MPL-001) — MPL-001: which is a 25:1 Cannabidiol (CBD): ∆9-tetrahydrocannabidiol (THC) oral formulation with a concentration of 50 mg/ml of CBD and 2 mg/ml of THC. The starting dose will be 1 mL per day (50 mg CBD) orally and gradually titrated to a maximum dose of 6 mL (300 mg CBD) per day in a divided dosage within 6 to 8 weeks of treatment initiation based on patient assessment. Once the optimal dose has been determined, which maximizes potential therapeutic effects while minimizing adverse effects, the dose will be maintained for the remainder of the trial.
  Other Names: CBD concentrate
  Arms: CBD oil
Drug: CDB+THC oil (MPL-005) — MPL-005: which is a 5:1 Cannabidiol (CBD):∆9-tetrahydrocannabidiol (THC) oral formulation with a concentration of 25 mg/ml of CBD and 5 mg/ml of THC. The starting dose will be 1 mL per day (25 mg CBD + 5 mg THC) orally and gradually titrated to a maximum dose of 6 mL (150 mg CBD + 30 mg THC) per day in a divided dosage within 6 to 8 weeks of treatment initiation based on patient assessment. Once the optimal dose has been determined, which maximizes potential therapeutic effects while minimizing adverse effects, the dose will be maintained for the remainder of the trial.
  Other Names: CBD concentrate
  Arms: CBD+THC oil
Drug: Placebo oil — The starting dose will be 1 mL per day (contains no API) orally and gradually titrated to a maximum dose of 6 mL per day in a divided dosage within 6 to 8 weeks of treatment initiation based on patient assessment. Once the optimal dose has been determined, which maximizes potential therapeutic effects while minimizing adverse effects, the dose will be maintained for the remainder of the trial.
  Other Names: Matching placebo
  Arms: Placebo oil

SUMMARY:
The investigators are conducting a pilot (i.e. a small study) in order to find out the effectiveness and safety of medical cannabis in the management of chronic pain. At the end of this 3 month study, investigators will gather information on how easy it is for patients to enroll and complete the entire study. The results of this pilot study will help the study team design a larger randomized controlled trial.

DETAILED DESCRIPTION:
Chronic pain is defined as pain lasting longer than three months, affects ~20% of Canadian adults. In addition to having a significant negative impact at the individual patient level (i.e., decreased quality of life and functioning), chronic pain is also a main cause of disability and health care use. Opioids are frequently prescribed to manage chronic pain despite limited data on their long term usefulness and has become one of the major contributors to the current opioid crisis in Canada. Chronic pain can potentially be treated with medical cannabis as an adjunct or alternative to opioids due to their similar behavioral, anatomical and biochemical mechanisms. Cannabinoids also potentially prevent the development of tolerance to opioids when co-administered.

Cannabinoids have demonstrated the ability to reduce pain as well as opioid-sparing effects in pre-clinical and clinical studies however further research is needed to identify the optimal make-up, ratio, and dosage of cannabinoids to minimize harms and maximize benefits. Furthermore, studies conducted to date have methodological problems such as short follow-up windows (hours or days) that limit conclusions. The investigators therefore propose a randomized, placebo-controlled trial of oral cannabinoids [CBD (cannabidiol) alone or in combination with THC (delta-9-tetrahydrocannabinol)] for reducing pain disability and opioid use for pain management in chronic pain. However, there are a number of feasibility issues that should be addressed prior to launching a full-scale trial in this area. Some issues have been identified in the literature (e.g., success of blinding) while others are related to the changing socio-medico-legal landscape surrounding cannabis use in Canada.

The purpose of this pilot study is to test the study plan, patient recruitment and compliance with the study procedures. Results of this study may be used as a guide for larger studies and will help us determine if medical cannabis can reduce daily opioid doses and/or decrease pain interference (disability) in chronic pain patients.

This study will aim to recruit 51 patients from the Toronto General Hospital Transitional Pain Service.

Study Procedure: After obtaining the Informed consent, patients will be randomized into one of the three study groups. Patients will either receive CBD oil, CBD+THC oil or placebo orally for 12 weeks. Starting dose will be 1 ml per day. The dose of study drug will be adjusted based on patients' reported efficacy and adverse effects. After starting the study drug, patients will have scheduled study visits either remotely or in-person at 4, 8, and 12 weeks plus a follow up calls or virtual clinic visit(OTN) at 2 and 6 weeks. At every study visit, patients will be asked to complete the questionnaires that will assess their pain level and how it affects their quality of life, opioid use, and side effects if they are experiencing. The investigators will also collect information on: demographic and baseline characteristics (e.g., sex, age, height, weight, and body mass index) and medical history (including prior and concomitant medications) via patient interview or from inspection of medical records. Additionally, symptoms of depression and anxiety will be measured with the validated screening tools at baseline and 12 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 25 years
2. Able to understand and read English
3. Experiencing chronic, non-palliative pain

Exclusion Criteria:

1. Use of nabilone, nabiximols or cannabis in the 30 days preceding study recruitment
2. Known allergy to cannabis or any cannabinoid
3. Serious ongoing medical issues (i.e., lung, liver, kidney or heart disease) that in the opinion of the Investigator would compromise the safety of the patient
4. Current uncontrolled serious mental disorders such as schizophrenia, or psychosis
5. Currently pregnant or breast-feeding (a negative urine pregnancy test must be obtained for women of child bearing potential during pretreatment evaluation)
6. Men and women planning to start a family in the next 12 weeks
7. Has declared a current alcohol or substance use disorder (excluding opioid use disorder)
8. Currently using Methadone or Buprenorphine
9. Patients who are naïve to pain treatments

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome: pertaining to the patients recruitment | Through study completion, an average of 1 year
  The ability to recruit the necessary number of patients during the estimated 12-month period
Feasibility outcome: pertaining to adherence to intervention | Up to 12 weeks post-treatment
  Defined as ≥70% of patients taking ≥70% of the prescribed doses and assessed from the participant-kept study drug diary data at each study visit.
Feasibility outcome: pertaining to withdrawal from study | Up to 12 weeks post-treatment
  Participant withdrawal from the study <20%
Feasibility outcome: pertaining to questionnaire data | Up to 12 weeks post-treatment
  The amount of missing data from all questionnaires <20%
Feasibility outcome: the rate of unintentional unblinding | Up to 12 weeks post-treatment
  Defined as the participant correctly identifying group allocation and blinding success will be quantified using the BANG Index.

SECONDARY OUTCOMES:
The mean Morphine Equivalent (MEQ) dose (mg/day) at 12 weeks post-treatment for patients that were consuming opioids at the start of the trial | Baseline and at 2-,4-,6-,8- and 12-weeks post-treatment
  The data for opioid consumption will be extracted from the medical record or obtained via self report. MEQ will be calculated based on the 2017 Canadian Guideline for Safe and Effective Use of Opioids for Chronic Non-Cancer Pain.
The mean pain interference at 12 weeks post-treatment | Baseline and at 2-,4-,6-,8- and 12-weeks post-treatment
  Pain interference will be assessed with The Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference - Short Form 8a scale. This validated scale consists of 8 items detailing the extent to which pain interferes with the individual's abilities to perform and enjoy daily life; each item is rated on a 5-point scale (1=not at all, 2=a little bit, 3=somewhat, 4=quite a bit and 5=very much). Scores are calculated from the total of item responses, with higher scores reflecting greater pain interference.

OTHER OUTCOMES:
The proportion of patients weaned off opioids at 12 weeks post-treatment initiation for patients that were consuming opioids at the start of the trial | 12-weeks post-treatment
  Defined as no opioid use on the day prior to the final study visit
Mean pain severity scores at 12-weeks post-treatment | Baseline and at 2-,4-,6-,8- and 12-weeks post-treatment
  Pain severity will be assessed with three separate numeric rating scales (NRS): pain now, pain at its maximum in the past 24 hours, and pain at its minimum in the past 24 hours. Each NRS will range from 0 "not at all severe" to 10 "pain as bad as you can imagine. Higher scores indicate greater pain severity.
Overall improvement related to the intervention | Baseline and at 2-,4-,6-,8- and 12-weeks post-treatment
  Overall improvement related to the intervention will be assessed with the Patient Global Impression of Change Scale (PGIC). PGIC is a single item rated on a 7-point scale from "very much improved" to "very much worse".
Adverse events assessment | Baseline and at 2-,4-,6-,8- and 12-weeks post-treatment
  Adverse events will be assessed with the Toronto Side Effects Scale (TSES), a measure of the incidence, frequency and severity of 31 adverse events plus an open-ended item.
Assessment of symptoms of anxiety | Baseline and at 12-weeks post-treatment
  The symptoms of anxiety will be measured using Generalized Anxiety Disorder 7-item scale (GAD-7). This 7-item scale assesses the signs of GAD (e.g. ''Feeling afraid as if something awful might happen") with response option of : 0= Not at all, 1=Several days, 2= More than half the days and 3= Nearly everyday. Scores are calculated from the total of item responses, with higher scores reflecting greater anxiety.
Assessment of symptoms of depression | Baseline and at 12-weeks post-treatment
  The symptoms of depression will be measured by Patient Health Questionnaire 9 item scale (PHQ-9).
  The PHQ-9 assesses the signs of depression (e.g. Little interest or pleasure in doing things) with response option of :
  0= Not at all, 1= Several days, 2= More than half the days, 3= Nearly everyday. Scores are calculated from the total of item responses, with higher scores reflecting the greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hance Clarke, MD, PhD, Principal Investigator — Toronto General Hospital, UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No